CLINICAL TRIAL: NCT04728776
Title: Translation and Validation of Stroke Impact Scale 3.0 in Urdu for Pakistan
Status: Completed | Type: Observational
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Other Study IDs: 293
Record Dates: First submitted 2021-01-20; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND Knowledge about the perceived impact of stroke on survivors' lives is still scarce in Pakistan due to the lack of translated and culturally adapted self-rating scales. The stroke impact scale is a comprehensive self-reported outcome measure designed to assess the quality of life following the stroke. Although the psychometric properties of SIS found to be superior to the conventional generic quality of life scales, it has not been translated and tested in Pakistan.

OBJECTIVE To translate and cross-culturally validate the Urdu version of stroke impact scale 3.0 for Pakistan MATERIAL AND METHODS Established guidelines were followed for translation and adaption of the Stroke impact scale 3.0. A prospective cohort of 116 patients with mild to moderate stroke self-reported their recovery on the Urdu version of SIS 3.0. The patients were concurrently evaluated on the established scales to assess the validity using the Spearman correlation coefficient. ANOVA was used to determine the discriminant validity. Ninety patients were consecutively re-evaluated to determine the test-retest reliability, precision, minimal detectable change (MCD) and clinically minimally important difference. The coefficients of ICC, Cronbach's alpha, and weighted kappa were calculated to establish the stability and consistency of the scale. The receiver operating curve was used to estimate the MCID of SIS-16 using global rating scale as an anchor.

KEYWORDS: Stroke, Stroke Impact Scale, Outcome Measures, Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute, subacute or chronic stroke
* Patients with hemorrhagic or ischemic or recurrent stroke attack
* Age of patients between 50-80
* Ability to read and write Urdu with minimum education to 5th grade

Exclusion Criteria:

* Patients with severe neurological comorbidities
* Patients having communication difficulties, such as patients with global aphasia or reduced consciousness.

Ages: 50 Years to 80 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute, subacute or chronic stroke-hemorrhagic or ischemic or recurrent stroke attack, age of patients between 50-80 and the ability to read and write Urdu with minimum education to 5th grade. Patients were not enrolled in the study if they presented with severe neurological comorbidities and communication difficulties, such as patients with global aphasia or reduced consciousness.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Stroke Impact Scale 3.0 "Change" is being assessed | Day 1, A week after the first assessment
  A 59-item self-reported scale with 8 domains, scores of each domain range from 0 to 100, and higher scores indicate a better health-related quality of life
Stroke Impact Scale-16 "Change" is being assessed | Day 1, A week after the first assessment and at discharge upto 12 weeks
  It consists of 16 items of 4 physical function. Its score varies from 0 to 100 and higher score indicates more functioning of the patient

SECONDARY OUTCOMES:
Short-form 36, "Change" is being assessed | Day 1, A week after the first assessment
  SF-36 is a generic HRQoL measure that includes 8 domains. Scores for each domain range from 0 to 100, and higher values indicate better function.
Barthel Index, "Change" is being assessed | Day 1, A week after the first assessment
  The Barthel Index used to evaluate activities of daily living in stroke patients measures and measures 10 basic aspects of activities of daily living related to self-care and mobility: control of bowels and bladder, grooming, toilet use, feeding, transfer, mobility, dressing, stairs, and bathing. Its score ranges from 0 to 100, and lower scores indicate greater dependency.
Stroke Rehabilitation Assessment of Movement, "Change" is being assessed | Day 1, A week after the first assessment
  Composed of 30 items, score range from 0-100, measures physical function and higher score indicates more physical functioning of patient
Modified Rivermead Mobility Index, "Change" is being assessed | Day 1, A week after the first assessment
  A 15-items scale with each item score range from 0 to 5. Its score varies from 0 to 100 and higher score indicates more functioning of the patient
Global rating of change scale "Change" is being assessed | at discharge up to 12 weeks only, Please note it simply ask the patient how much change he has experienced over the course of treatment period
  Measures self-perceived change in health status and the main purpose is to quantify the extent to which a patient has improved or deteriorated over time. Score lower than 0 means patient has deteriorated and more than 0 means patient has improved. Its score varies from -7 to +7

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale, "Change" is being assessed | Day 1, A week after the first assessment, at discharge upto 12 week
  The Hospital Anxiety and Depression Scale is 14 items scale for assessment of anxiety and depression. Scale consists of 7 items for depression and 7 items for depression and each item scored from 0 (no problem) to 3 (severe problem). Scores on individual items can be summed to calculate a score for anxiety and for depression and higher score is indicative of more depression and anxiety. Score of each sub scale varies from 0-21, where 0-7 means normal, 8-10 means mild, 11-14 means moderate, 15-21 means sever disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- The University Of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan